CLINICAL TRIAL: NCT06549686
Title: A Phase III Study Evaluating the Efficacy and Safety of CLS2901C in Patients With Osteoarthritis of the Knee
Brief Title: A Phase III Study of CLS2901C in Patients With Osteoarthritis of the Knee
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CellSeed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLS2901-OAK-01
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the osteotomy monotherapy group (No Intervention): the osteotomy monotherapy
- the osteotomy + RMSC combination therapy group (Experimental): the osteotomy + RMSC combination therapy
  *RMSC combination therapy R: Resection of unhealthy tissue MS: Marrow arrow Stimulating＝MSCs Recruitment C: Covered by Chondrocyte sheets
  Interventions: Biological: CLS2901C (human [allogeneic] chondrocyte sheets)

INTERVENTIONS:
Biological: CLS2901C (human [allogeneic] chondrocyte sheets) — CLS2901C (human [allogeneic] chondrocyte sheets)
  Arms: the osteotomy + RMSC combination therapy group

SUMMARY:
To evaluate the efficacy and safety of CLS2901C human allogenic chondrocyte sheets used in the osteotomy + RMSC group compared to in the osteotomy alone group of patients with osteoarthritis of the knee (OAK).

DETAILED DESCRIPTION:
The investigational human cellular based product is a cell sheet made by culturing and growing chondrocytes taken from cartilage tissue derived from patients with polydactyly. To evaluate the efficacy and safety of CLS2901C human allogenic chondrocyte sheets used in the osteotomy + RMSC group compared to in the osteotomy alone group of patients with osteoarthritis of the knee (OAK). Safety is evaluated by the rate of adverse events and malfunctions. The evaluation period for each group will be approximately 14.5 months, and after the completion of the 52-week evaluation, patients who are available for follow-up will continue to be examined and observed for 5 years after sheets transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 20 to 79 years at informed consent.
2. Diagnosis of OAK classified as Kellgren-Lawrence (K-L) Grade 2 to 4 based on plain lower extremity X-ray.
3. OAK eligible for proximal tibial osteotomy based on the following criteria: Range of motion (ROM): >=120 degree flexion, <=5 degree extension
4. Preoperative cartilage defect of the femoral condyle/trochlear groove or medial tibial condyle with an area of >=4 cm2 per defect site.
5. Total defect area of <=21 cm2 in individuals with multiple cartilage defects.
6. Body mass index (BMI) <30.
7. No coexisting ligament injury requiring surgery, and no meniscal injury requiring suturing or surgical repair other than partial resection, in the target knee.
8. No history of ligament reconstruction, meniscal suturing, total meniscectomy or bone marrow stimulation, and no history of treatment with regenerative medicine products (including investigational products), cell processing products or gene therapy, in the target knee.
9. No history of treatment with hyaluronic acid products and/or opioid for severe pain in the target knee within 1 month prior to informed consent.
10. No history of treatment with corticosteroid products and/or immunosuppressive drug in the target knee within 3 months prior to informed consent.
11. No history of platelet-rich plasma (PRP) therapy within 6 months prior to informed consent.
12. Non-smoker; provided, however, that smokers will be eligible for study entry if they consent to abstain from smoking from 3 months prior to proximal tibial osteotomy or proximal tibial osteotomy+RMSC until postoperative bone healing.
13. Written informed consent to participate in the study on a voluntary basis.

Exclusion Criteria:

1. Requires surgical treatment of the non-target knee during the study period.
2. Any coexisting illness that would interfere with surgery under general anesthesia or that would affect knee surgery.
3. Systemic inflammatory disease such as rheumatoid arthritis.
4. Systemic Active infectious disease such as bacterial, fungal or viral infection.

6) Serious disease such as liver disorder, renal disorder, heart disease, lung disease, blood disease or metabolic disease that would make the patient unsuitable for study entry in the opinion of the investigator.

7) Diagnosed or suspected malignant tumor or history of malignant tumor within the past 5 years.

8) Uncontrolled psychiatric disorder. 9) Poorly-controlled diabetes (HbA1c: >7.0%). 10) septic arthritis of the target knee. 11) Women who are pregnant or breastfeeding, or women of childbearing potential. Women of childbearing potential must agree to use the following contraceptive methods (i.e., contraceptives and medical devices that are approved/certified in Japan) or to abstain completely from sexual intercourse from the time of informed consent and for the study duration (excluding the follow-up period) in order to be eligible for study entry. (a) Primary contraceptive methods: Oral contraceptives, intrauterine devices (IUDs) including progesterone-releasing systems. (b) Adjunctive contraceptive methods: Condoms Use of a primary contraceptive method is mandatory, whereas use of the adjunctive contraceptive method must be in conjunction with a primary contraceptive method. Given that oral contraceptive doses can be missed and that their effects may be diminished when used concomitantly with other medications or dietary health supplements, subjects should consider changing their primary contraceptive method.

12) Participated in another clinical study within the past 6 months, currently participating in another clinical study, or planning to participate in another clinical study while also participating in the present study.

13) Known history of hypersensitivity to antibiotics (benzylpenicillin potassium, streptomycin sulfate, amphotericin B).

14) Known history of hypersensitivity to bovine-derived materials. 15) Any other reason the investigator deems the subject unsuitable for study entry.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
KOOS 4 score (The Knee injury and Osteoarthritis Outcome 4 score) | 52 weeks
  Absolute change from baseline KOOS4 (Pain, Symptoms, ADL, QOL) score at postoperative Week 52. The four patient-relevant subscales of KOOS are scored separately: KOOS Pain (9items); KOOS Symptoms (7 items); KOOS ADL (17 items); KOOS QOL (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as is common in orthopaedic assessment scales and generic measures.

CONTACTS AND LOCATIONS:
Overall Officials: Manabu Ishizuka, Study Director — CellSeed Inc.
Locations (6):
- Japan (6):
  - Ebina General Hospital/Ebina Medical Plaza, Ebina, Kanagawa
  - Tokai University Hospital, Isehara, Kanagawa
  - Yokohama Sekishinkai Hospital, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokohama Minami Kyousai Hospital, Yokohama, Kanagawa
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No